CLINICAL TRIAL: NCT04898166
Title: Association of Androgenetic Alopecia and Severity of Coronavirus Disease 2019 (COVID-19)
Status: Completed | Type: Observational
Sponsor: Syeda Mahanum Ali (Other Government)
Responsible Party: Sponsor-Investigator, Syeda Mahanum Ali, Postgraduate trainee dermatology, Jinnah Postgraduate Medical Centre
Organization: Jinnah Postgraduate Medical Centre (Other Government)
Other Study IDs: NO.F.2-81/2021-GEN/56923/JPMC
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Androgenetic Alopecia; Coronavirus Disease 2019; Covid19; Male Pattern Baldness; Female Pattern Baldness; COVID-19 Pneumonia
Keywords: Covid19; Androgenetic alopecia
MeSH Terms: conditions — Alopecia; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) can cause variable symptoms ranging from mild common cold-like symptoms to severe life threatening pneumonia. Recent studies show severe outcomes of COVID-19 patients specially in males who suffer from androgenetic alopecia, would be significant and is of particular interest of this study and could help further support the hypothesis that anti-androgen therapy might represents an additional potential intervention against severe COVID-19.

DETAILED DESCRIPTION:
INTRODUCTION: An outbreak of Corona virus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-coV-2) occurred in Wuhan city, Hubei province, China in December 2019. Belonging to the family Beta-coronavirus, this virus can cause variable symptoms ranging from mild common cold-like symptoms to severe life threatening pneumonia. Numerous cases of new onset of skin lesions in COVID-19 patients are spreading across the globe. There are also some reports of aggravation of prior skin disorders. While severe COVID-19 symptoms and high mortality primarily manifested in older adults specially adult males, this sexual dimorphism in the severity of COVID-19 patients predisposed possibly due to increased androgen levels particularly in males suffering from androgenetic alopecia (AGA) would be significant and is of particular interest of this study and could help further support the hypothesis that anti-androgen therapy might represents an additional potential intervention against severe COVID-19.

OBJECTIVE: Association of Androgenetic alopecia and severity of Coronavirus disease 2019 (COVID-19).

PLACE OF STUDY: COVID-19 isolation unit of Jinnah postgraduate medical center (JPMC) Karachi, Sindh province, Pakistan.

RESEARCH METHODOLOGY: This study will be conducted on patients admitted in COVID-19 isolation unit of JPMC Karachi. Permission from the institutional ethical review committee will be taken prior to conduction of study, demographic data and written informed consent will be taken from every patient. Sample size of study would be 300 hospitalized patients of COVID-19. Detailed history and examination of patients including be conducted in COVID-19 patients. Scoring of AGA be evaluated using Hamilton-Norwood scale (HNS) in men and Ludwig scale in female. Severity of the COVID-19 be measured by COVID severity score (A-DROP). Study is aimed to evaluate association of AGA and severity of COVID-19, frequency of AGA in covid 19 and whether the lung involvement correlates with the severity of AGA or whether the proportion of AGA is higher in intensive care/fatal COVID-19.

DATA ANALYSIS: Data will be analysed using SPSS version 23 registered for Microsoft windows. Mean and standard deviation will be calculated for expression of quantitative variables like age, weight, duration of disease symptoms. Frequencies and percentages will be calculated for the qualitative variables like gender, co-morbidities, frequency and severity of AGA, disease outcome and AGA associated with severity of COVID-19. Effect modifiers like age, gender, weight, co-morbidities, duration of symptoms will be controlled through stratification. Post-stratification will be recalculated and chi-square test will be applied. P-value of <0.05% will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients of diagnosed covid-19 age > 20years
* with or without androgenetic alopecia
* with or without comorbidities
* irrespective of disease duration -

Exclusion Criteria:

* none

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalised diagnosed covid-19 patients with or without comorbidities. Irrespective of disease duration. Intensity and frequency of androgenetic alopecia, disease outcome be noted in these patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, MBBS, FCPS, SCE-Derm(MRCP-UK), Principal Investigator — Jinnah Postgraduate Medical Centre; Syeda Mahanum Ali, MBBS, Postgraduate Trainee, Principal Investigator — Jinnah Postgraduate Medical Centre
Locations (1):
- Jinnah postgraduate medical center, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Goren A, McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Dhurat R, Washenik K, Lotti T. What does androgenetic alopecia have to do with COVID-19? An insight into a potential new therapy. Dermatol Ther. 2020 Jul;33(4):e13365. doi: 10.1111/dth.13365. Epub 2020 Apr 8. No abstract available. PMID 32237190
- [Background] Muller Ramos P, Ianhez M, Amante Miot H. Alopecia and grey hair are associated with COVID-19 Severity. Exp Dermatol. 2020 Dec;29(12):1250-1252. doi: 10.1111/exd.14220. Epub 2020 Nov 18. No abstract available. PMID 33098701
- [Background] Goren A, Vano-Galvan S, Wambier CG, McCoy J, Gomez-Zubiaur A, Moreno-Arrones OM, Shapiro J, Sinclair RD, Gold MH, Kovacevic M, Mesinkovska NA, Goldust M, Washenik K. A preliminary observation: Male pattern hair loss among hospitalized COVID-19 patients in Spain - A potential clue to the role of androgens in COVID-19 severity. J Cosmet Dermatol. 2020 Jul;19(7):1545-1547. doi: 10.1111/jocd.13443. Epub 2020 Apr 23. PMID 32301221
- [Background] Wambier CG, Vano-Galvan S, McCoy J, Gomez-Zubiaur A, Herrera S, Hermosa-Gelbard A, Moreno-Arrones OM, Jimenez-Gomez N, Gonzalez-Cantero A, Fonda-Pascual P, Segurado-Miravalles G, Shapiro J, Perez-Garcia B, Goren A. Androgenetic alopecia present in the majority of patients hospitalized with COVID-19: The "Gabrin sign". J Am Acad Dermatol. 2020 Aug;83(2):680-682. doi: 10.1016/j.jaad.2020.05.079. Epub 2020 May 22. PMID 32446821
- [Background] McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Sinclair R, Ramos PM, Washenik K, Andrade M, Herrera S, Goren A. Racial variations in COVID-19 deaths may be due to androgen receptor genetic variants associated with prostate cancer and androgenetic alopecia. Are anti-androgens a potential treatment for COVID-19? J Cosmet Dermatol. 2020 Jul;19(7):1542-1543. doi: 10.1111/jocd.13455. Epub 2020 Jun 14. No abstract available. PMID 32333494
- [Background] Lee J, Yousaf A, Fang W, Kolodney MS. Male balding is a major risk factor for severe COVID-19. J Am Acad Dermatol. 2020 Nov;83(5):e353-e354. doi: 10.1016/j.jaad.2020.07.062. Epub 2020 Jul 22. PMID 32707256
- [Background] Wambier CG, Vano-Galvan S, McCoy J, Pai S, Dhurat R, Goren A. Androgenetic alopecia in COVID-19: Compared to age-matched epidemiologic studies and hospital outcomes with or without the Gabrin sign. J Am Acad Dermatol. 2020 Dec;83(6):e453-e454. doi: 10.1016/j.jaad.2020.07.099. Epub 2020 Jul 29. PMID 32735970
- See also: What does androgenetic alopecia have to do with COVID-19? An insight into a potential new therapy — https://pubmed.ncbi.nlm.nih.gov/32237190/
- See also: Alopecia and grey hair are associated with COVID-19 Severity — https://pubmed.ncbi.nlm.nih.gov/33098701/
- See also: A preliminary observation: Male pattern hair loss among hospitalized COVID-19 patients in Spain - A potential clue to the role of androgens in COVID-19 severity — https://pubmed.ncbi.nlm.nih.gov/32301221/
- See also: Androgenetic alopecia present in the majority of patients hospitalized with COVID-19: The "Gabrin sign" — https://pubmed.ncbi.nlm.nih.gov/32446821/
- See also: Racial variations in COVID-19 deaths may be due to androgen receptor genetic variants associated with prostate cancer and androgenetic alopecia. Are anti-androgens a potential treatment for COVID-19? — https://pubmed.ncbi.nlm.nih.gov/32333494/
- See also: Male balding is a major risk factor for severe COVID-19 — https://pubmed.ncbi.nlm.nih.gov/32707256/
- See also: Androgenetic alopecia in COVID-19: Compared to age-matched epidemiologic studies and hospital outcomes with or without the Gabrin sign — https://pubmed.ncbi.nlm.nih.gov/32735970/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 300 participants at COVID-19 isolation unit jinnah postgraduate medical centre karachi.
Pre-assignment Details: * 300 participants signed consent for participation.
  * 300 participants assigned for the study.
Groups:
- 220 Hospitalized Male Participants Diagnosed Case of COVID-19.: 220 hospitalised male participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
- 80 Hospitalized Female Participants Diagnosed Case of COVID-19.: 80 hospitalized female Participants diagnosed case of hospitalized COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught ludwig scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
Period: Overall Study
Arm/Group | 220 Hospitalized Male Participants Diagnosed Case of COVID-19. | 80 Hospitalized Female Participants Diagnosed Case of COVID-19.
Started | 220 | 80
Completed | 220 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 220 Hospitalized Male Participants Diagnosed Case of COVID-19.: 220 hospitalized male Participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
- 80 Hospitalized Female Participants Diagnosed Case of COVID-19: 80 hospitalized female Participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught ludwig scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
- Total: Total of all reporting groups
Arm/Group | 220 Hospitalized Male Participants Diagnosed Case of COVID-19. | 80 Hospitalized Female Participants Diagnosed Case of COVID-19 | Total
Number analyzed (Participants) | 220 | 80 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.39 (14.928) | 52.17 (8.391) | 53.06 (13.5)
Age, Customized [Count of Participants; unit: Participants]
  Between 20 to 40 years | 41 | 29 | 70
  Between >40 to 60 years | 99 | 51 | 150
  >60 years | 80 | 00 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 00 | 80 | 80
  Male | 220 | 00 | 220
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 00 | 00 | 0
  Not Hispanic or Latino | 220 | 80 | 300
  Unknown or Not Reported | 00 | 00 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 220 | 80 | 300
Comorbidities [Count of Participants; unit: Participants]
  Smoking | 14 | 2 | 16
  Ischemic heart disease | 12 | 4 | 16
  Diabetes mellitus | 35 | 17 | 52
  Hypertension | 34 | 17 | 51
  Obesity | 15 | 6 | 21
  Chronic kidney disease | 10 | 5 | 15
  Multiple comorbidities | 20 | 19 | 39
  No comorbidity | 82 | 10 | 92

OUTCOME MEASURES:

1. Primary Outcome: Androgenetic Alopecia Frequency in Participants.
Description: Frequency of Androgenetic alopecia in patients be noted.
Time Frame: Day 1 of admission
Measure: Count of Participants; unit: Participants
Groups:
- 220 Hospitalized Participants Diagnosed Case of COVID-19.: 220 hospitalised male participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
- 80 Hospitalized Female Participants Diagnosed Case of Hospitalized COVID-19: 80 hospitalized female Participants diagnosed case of hospitalized COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught ludwig scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
Arm/Group | 220 Hospitalized Participants Diagnosed Case of COVID-19. | 80 Hospitalized Female Participants Diagnosed Case of Hospitalized COVID-19
Number analyzed (Participants) | 220 | 80
Participants
  With androgenetic alopecia | 209 | 37
  Without androgenetic alopecia | 11 | 43

2. Primary Outcome: Severity of Androgenetic Alopecia in Patients
Description: Severity of androgenetic alopecia be measured using Hamilton and norwood scale (HNS) less than 3 or 3-7.
  In females using ludwig scale: less than 2 or 2-3. Hamilton norwood score: Minimum value 1, maximum value 7. Ludwig score: minimum 0, maximum 3 Mild to moderate: HNS <3/ Ludwig <2 Severe: HNS 3-7/ ludwig 2-3
Time Frame: Day 1 of admission
Measure: Count of Participants; unit: Participants
Groups:
- 220 Hospitalised Male Participants Diagnosed Case of COVID-19.: 220 hospitalised male participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
Arm/Group | 220 Hospitalised Male Participants Diagnosed Case of COVID-19. | 80 Hospitalized Female Participants Diagnosed Case of Hospitalized COVID-19.
Number analyzed (Participants) | 220 | 37
Participants
  Mild to moderate | 43 | 9
  Severe | 177 | 28

3. Primary Outcome: 300 Participants Mean Age
Description: Age of the patient is very important to co-relate with disease outcome and severity of Androgenetic alopecia
Time Frame: Day 1 of admission
Measure: Mean (Standard Deviation); unit: years
Groups:
- 300 Participants Diagnosed Case of Hospitalized COVID-19. Mean Age be Noted: 300 Participants diagnosed case of hospitalized COVID-19. Mean age be noted in both males and females
Arm/Group | 300 Participants Diagnosed Case of Hospitalized COVID-19. Mean Age be Noted
Number analyzed (Participants) | 300
years | 53.06 (13.495)

4. Primary Outcome: Disease Outcome as Assessed by Number of Participants Experiencing Better or Worst Outcome With Respect to Age Group.
Description: Outcome of participants suffering from covid-19 with respect to age group as better outcomes: oxygen mask/bag or nasal cannula Worst outcomes: ventilator or death
Time Frame: From date of randomization until the date of clinical improvement (discharge, from ventilator to mask/nasal cannula) or worsening of condtion(from mask/bag to ventilator) or death from any cause, assessed up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | 220 Hospitalised Male Participants Diagnosed Case of COVID-19. | 80 Hospitalized Female Participants Diagnosed Case of Hospitalized COVID-19.
Number analyzed (Participants) | 220 | 80
Participants
  Participants on mask/bag with age 20-40years | 15 | 10
  Participants on mask/bag with age >40-60 years | 13 | 18
  Participants on mask/bag with age >60years | 13 | 0
  Participants on Nasal cannula with age 20-40years | 15 | 4
  Participants on nasal cannula with age >40-60 years | 37 | 12
  Participants on nasal cannula with age >60years | 20 | 0
  Participants on ventilator with age 20-40years | 4 | 11
  Participants on ventilator with age >40-60 years | 16 | 15
  Participants on ventilator with age >60years | 10 | 0
  Participants death with age 20-40 years | 7 | 4
  Participants death with age >40-60 years | 33 | 6
  Participants death with age >60years | 37 | 0

5. Primary Outcome: Disease Outcome as Assessed by Severity of Androgeneic Alopecia in Males
Description: Covid-19 disease outcome assessed by Severity of androgenetic alopecia to find out their correlation
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- 220 Hospitalised Male Subjects. Their Disease Outcomes in Relation to Severity of AGA: 220 hospitalised male participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of Androgenetic alopecia be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death. Their disease outcomes in relation to severity of AGA
Arm/Group | 220 Hospitalised Male Subjects. Their Disease Outcomes in Relation to Severity of AGA
Number analyzed (Participants) | 220
Participants
  Patients on nasal cannula with HNS <3 | 20
  Patients on nasal cannula with HNS 3-7 | 52
  Patients on mask/bag with HNS <3 | 14
  Patients on mask/bag with HNS 3-7 | 27
  Patients on ventilator with HNS <3 | 5
  Patients on ventilator with HNS 3-7 | 25
  Patients death with HNS <3 | 4
  Patients death with HNS 3-7 | 73
Statistical Analysis 1: Comparison: 220 Hospitalised Male Subjects. Their Disease Outcomes in Relation to Severity of AGA; Test type: Superiority; p = 0.000, Chi-squared; Chi-square value 18.90 and its asymptotic significance .000

6. Primary Outcome: Disease Outcome be Assessed by Severity of Androgenetic Alopecia in Females
Description: Covid-19 disease outcome assessed by Severity of androgenetic alopecia to find out their correlation
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- 80 Hospitalised Female Participants. Their Disease Outcomes in Relation to Severity of AGA: 80 hospitalised female participants diagnosed case of COVID-19. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught ludwig scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death. Their disease outcomes in relation to severity of AGA
Arm/Group | 80 Hospitalised Female Participants. Their Disease Outcomes in Relation to Severity of AGA
Number analyzed (Participants) | 80
Participants
  Female participants on mask/bag with no androgenetic alopecia | 9
  Female participants on mask/bag with ludwig scale <2 | 3
  Female participants on mask/bag with ludwig scale 2-3 | 4
  Female participants on nasal cannula without androgenetic alopecia | 17
  Female participants on nasal cannula with ludwig scale <2 | 3
  Female participants on nasal cannula with ludwig scale 2-3 | 8
  Female participants on ventilator with no androgenetic alopecia | 14
  Female participants on ventilator with ludwig scale <2 | 3
  Female participants on ventilator with ludwig scale 2-3 | 9
  Female participants death with no androgenetic alopecia | 3
  Female participants death with ludwig scale <2 | 0
  Female participants death with ludwig scale 2-3 | 7
Statistical Analysis 1: Comparison: 80 Hospitalised Female Participants. Their Disease Outcomes in Relation to Severity of AGA; Test type: Superiority; p = 0.081, Chi-squared; Chi-square value 7.544 and its asymptotic significance .273

7. Primary Outcome: Covid-19 Disease Outcomes Correlating With Severity of Androgenetic Alopecia and Age in Females.
Description: It is to find out how severily disease outcomes can be affected due to androgeneic alopecia by age accordingly.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- 37 Hospitalised Female Participants of COVID-19 With Androgenetic Alopecia: 37 hospitalised female participants diagnosed case of COVID-19 presence of absence of androgenetic alopecia influencing outcome be noted as patient on mask/bag, nasal cannula, ventilator or death with respec to aget
- 43 Hospitalised Female Participants of COVID-19 Without Androgenetic Alopecia With Respect to Age: 43 hospitalised female participants diagnosed case of COVID-19 with androgenetic alopecia. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death with respect to age
Arm/Group | 37 Hospitalised Female Participants of COVID-19 With Androgenetic Alopecia | 43 Hospitalised Female Participants of COVID-19 Without Androgenetic Alopecia With Respect to Age
Number analyzed (Participants) | 37 | 43
Participants
  Age 20-40yrs: nasal cannula | 0 | 4
  Age >40-60yrs: nasal cannula | 7 | 5
  Age >60yrs nasal cannula | 00 | 00
  Age 20-40yrs: mask/bag | 3 | 7
  Age >40-60yrs: mask/bag | 8 | 10
  Age >60yrs mask/bag | 00 | 00
  Age 20-40yrs: ventilator | 6 | 5
  Age >40-60yrs: ventilator | 6 | 9
  Age >60yrs: ventilator | 00 | 00
  Age 20-40yrs: death | 3 | 1
  Age >40-60yrs: death | 4 | 2
  Age >60yrs: death | 00 | 00

8. Primary Outcome: Covid-19 Disease Outcomes Correlating With Severity of Androgenetic Alopecia and Age in Males
Description: It is to find out how severily disease outcomes can be affected due to androgeneic alopecia by age accordingly.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- 43 Hospitalised Male Participants Diagnosed Case of COVID-19 With HNS <3.: 43 hospitalised male participants diagnosed case of COVID-19 with HNS <3. Presence or absence of androgenetic alopecia be noted. Severity of androgeneic be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death with respect to age
- 177 Hospitalised Male Participants Diagnosed Case of COVID-19 With HNS >3-7: 177 hospitalised male participants diagnosed case of COVID-19 with HNS 3-7. Severity of androgeneic be noted throught Hamilton norwood scale. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death with respect to age
Arm/Group | 43 Hospitalised Male Participants Diagnosed Case of COVID-19 With HNS <3. | 177 Hospitalised Male Participants Diagnosed Case of COVID-19 With HNS >3-7
Number analyzed (Participants) | 43 | 177
Participants
  Nasal cannula Age 20-40yrs | 4 | 11
  Nasal cannula age >40-60yrs | 10 | 27
  Nasal cannula age >60yrs | 6 | 14
  Mask/bag age 20-40yrs | 6 | 9
  Mask/bag age >40-60yrs | 5 | 8
  Mask/bag age >60yrs | 3 | 10
  Ventilator age 20-40yrs | 1 | 3
  Ventilator age >40-60yrs | 2 | 14
  Ventilator age >60yr | 2 | 8
  Death age 20-40yrs | 0 | 7
  Death age >40-60yrs | 1 | 32
  Death age >60yrs | 3 | 34

9. Primary Outcome: Hospital Disease Outcome in 300 Subjects. Having 220 Males and 80 Females
Description: Hospital disease outcome as mask, cannnula, ventilator or death in 300 subjects. Having 220 males and 80 Females
Time Frame: Disease outcome during this 4 month duration of study.
Measure: Count of Participants; unit: Participants
Groups:
- 220 Hospitalized Participants Diagnosed Case of COVID-19.: 220 hospitalised male participants diagnosed case of COVID-19. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
- 80 Hospitalized Female Participants Diagnosed Case of Hospitalized COVID-19: 80 hospitalized female Participants diagnosed case of hospitalized COVID-19. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
Arm/Group | 220 Hospitalized Participants Diagnosed Case of COVID-19. | 80 Hospitalized Female Participants Diagnosed Case of Hospitalized COVID-19
Number analyzed (Participants) | 220 | 80
Participants
  Mask/bag | 41 | 28
  Nasal cannula | 72 | 16
  Ventilator usage | 30 | 26
  Death | 77 | 10

10. Secondary Outcome: Comorbidities Including Diabetes Mellitus, Smoking, Hypertension, Ischemic Heart Disease, Chronic Kidney Disease, Obesity in Participants
Description: Comorbidities in patients suffering from covid-19 is of great value as it affects disease outcome.number of patients suffrring from comorbidities eg: diabetes mellitus, smoking, hypertension, ischemic heart disease, chronic kidney disease, obesity.
Time Frame: Date of randomization until upto 4 months
Measure: Count of Participants; unit: Participants
Groups:
- 300 Participants Diagnosed Case of Hospitalized COVID-19 Outcome in Relation to Comorbidities: 300 Participants diagnosed case of hospitalized COVID-19. 220 males and 80 females. Presence or absence of comorbidities. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
Arm/Group | 300 Participants Diagnosed Case of Hospitalized COVID-19 Outcome in Relation to Comorbidities
Number analyzed (Participants) | 300
Participants
  participant on nasal cannula with no comorbidity | 29
  participant on nasal cannula with history of smoking | 6
  participant on nasal cannula with history of ischemic heart disease | 4
  participant on nasal cannula with history of diabetes mellitus | 12
  participant on nasal cannula with history of hypertension | 15
  participant on nasal cannula with history of obesity | 8
  participant on nasal cannula with history of chronic kidney disease | 5
  participant on nasal cannula with history of multiple comorbidities | 9
  participant on mask/bag with no comorbidity | 20
  Participants on mask/bag with history of smoking | 6
  participant on mask/bag with history of history of ischemic heart disease | 1
  participant on mask/bag with history of diabetes mellitus | 15
  participant on mask/bag with history of hypertension | 8
  participant on mask/bag with obesity | 6
  participant on mask/bag with history of chronic kidney disease | 4
  participant on mask/bag with history of multiple comorbidities | 9
  participant on ventilator with no comorbidity | 17
  Participants on Ventilator with history of smoking | 1
  participant on ventilator with history of ischemic heart disease | 2
  participant on ventilator with history of diabetes mellitus | 7
  participant on ventilator with history of hypertension | 10
  participant on ventilator with history of obesity | 6
  participant on Ventilator with history of chronic kidney disease | 1
  participant on ventilator with history of multiple comorbidities | 12
  Participants death with no comorbidity | 26
  participant death with history of smoking | 1
  participant death: history of ischemic heart disease | 9
  participant death with history diabetes mellitus | 18
  participant death with history of hypertension | 18
  participant death with history of obesity | 1
  participant death with history of kidney disease | 5
  participant death with history of multiple comorbidities | 9

11. Secondary Outcome: Disease Duration of COVID-19
Description: Duration of symptoms patients experiencing from the onset of symptoms till outcome.
Time Frame: Day 1 of admission, till disease outcome in upto 4 months
Measure: Mean (Standard Deviation); unit: Days
Groups:
- 300 Participants Diagnosed Case of Hospitalized COVID-19 Disease Duration: 300 Participants diagnosed case of hospitalized COVID-19 mean and standard deviation of disease duration.
Arm/Group | 300 Participants Diagnosed Case of Hospitalized COVID-19 Disease Duration
Number analyzed (Participants) | 300
Days | 11.79 (5.727)

ADVERSE EVENTS:
Time Frame: From date of randomization until the date of clinical improvement (discharge, from ventilator to mask/nasal cannula) or worsening of condition(from mask/bag to ventilator) or death from any cause, assessed up to 4 months
Description: Our participants are hospitalized COVID-19 patients. Their adverse events are categorised as on oxygen mask/bag,nasal cannula, ventilator or death.
  Other non serious adverse events are zero because all of our participants were having covid19 so they faced it's symptom and no any other adverse event separately
Groups:
- 300 Participants Diagnosed Case of Hospitalized COVID-19 With or Without Androgenetic Alopecia.: 300 Participants diagnosed case of hospitalized COVID-19. 220 males and 80 females. Presence or absence of androgenetic alopecia be noted in males and females. Severity of androgeneic throught be noted throught Hamilton norwood score and ludwig score, respectively. Severity of COVID-19 and outcome be noted as patient on mask/bag, nasal cannula, ventilator or death.
Arm/Group | 300 Participants Diagnosed Case of Hospitalized COVID-19 With or Without Androgenetic Alopecia.
All-Cause Mortality (participants affected / at risk) | 87/300
Serious Adverse Events (participants affected / at risk) | 300/300
Other Adverse Events (participants affected / at risk) | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 Participants Diagnosed Case of Hospitalized COVID-19 With or Without Androgenetic Alopecia. (N=300)
87 male and female participants death (Infections and infestations) | 87
Male and female participants on ventilator (Infections and infestations) | 56
Male and female participants on oxygen mask/bag (Infections and infestations) | 69
Male and female participants on nasal cannula (Infections and infestations) | 88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT04898166/Prot_SAP_000.pdf